CLINICAL TRIAL: NCT05570669
Title: Evaluation of Two Different Regimens of Colon Preparations for Advanced Cleaning Using a 2lt PEG-CS With Simethicone: a Randomized Controlled Study.
Brief Title: Evaluation of Two Different Regimens of Colon Preparations for Advanced Cleaning.
Acronym: ERACLES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Societa Italiana di Endoscopia Digestiva (Other)
Collaborators: Presidio Ospedaliero Sant Ottone Frangipane Avellino (Unknown); Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other); Azienda Policlinico Umberto I (Other); Ospedale di Manerbio ASST Garda (Unknown); Ospedale Civile San Giovanni di Dio Crotone (Unknown); Ospedale di Baggiovara Modena (Unknown); Ospedale S. Jacopo Pistoia (Unknown); Ospedale S. Martino Belluno (Unknown); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Federico II University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: ERACLES01/2020
Record Dates: First submitted 2022-09-27; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Colonoscopy
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Intervention Model Description: two groups randomized 1:1
Who Masked: Outcomes Assessor
Masking Description: the endoscopist analyzes the results and evaluates the cleaning without knowing the treatment followed by the patient
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- full dose (Experimental): Group A "delayed full-dose" regimen (study arm): intake of two large A sachets and 2 small B sachets from 20:30 to 22:00 the evening before the exam. Taking the remaining 2 envelopes A large e 2 small B envelopes from 10.30 pm to midnight the evening before the exam.
  Interventions: Drug: (Macrogol 4000 52,500 g + Sodium sulphate anhydrous 3,750 g + Simethicone 0,080 g) full dose
- split dose (Other): Group B "split-dose" regimen (control arm): intake of two large A sachets and two small B sachets from 20.30 to 22:00 the evening before the exam. The remaining two large A envelopes and two small B envelopes will be taken 5 hours earlier than the time when the exam is scheduled on the same day as the exam.
  Interventions: Drug: (Macrogol 4000 52,500 g + Sodium sulphate anhydrous 3,750 g + Simethicone 0,080 g) split dose

INTERVENTIONS:
Drug: (Macrogol 4000 52,500 g + Sodium sulphate anhydrous 3,750 g + Simethicone 0,080 g) full dose — Taking the colonoscopy preparation drug (Clensia) in a single administration
  Other Names: Clensia in full dose
  Arms: full dose
Drug: (Macrogol 4000 52,500 g + Sodium sulphate anhydrous 3,750 g + Simethicone 0,080 g) split dose — Taking the colonoscopy preparation drug (Clensia) in two stages of administration
  Other Names: Clensia in Split dose
  Arms: split dose

SUMMARY:
Multicenter, prospective, randomized, checked, open label, with blind evaluation, for compare the intestinal cleansing effectiveness of the regimen full-dose delayed (A) of Clensia vs split regimen (B) of Clensia, in patients undergoing endoscopy.

DETAILED DESCRIPTION:
Enrolled patients, after providing written informed consent, are randomized to the CLENSIA preparation scheme, delayed full-dose or split-dose regimen. The delayed full-dose regimen will constitute study arm A while the split-dose regimen will constitute the control arm B.

Participants will follow a slag-free diet in the three days preceding the colonoscopy (reduction in the consumption of fruit, vegetables and legumes). On the day before the colonoscopy, patients will be able to have a normal breakfast and lunch that are both free of fiber. The dietary indications will be delivered in writing to the patient by the health staff of the center involved in the trial. From the moment the preparation begins with the intake of the product, the intake of solid foods will no longer be allowed while clear liquids of the patient's choice can be taken freely up to two hours before the colonoscopy.

The study ends for each patient with the execution of each procedure / examination planned for the visit 2 The effectiveness of the preparation in terms of intestinal cleansing is assessed blindly (by the endoscopist) using the scale (Boston Bowel Preparation Scale).

ELIGIBILITY:
Inclusion Criteria:

* Male / female patients
* outpatient, consecutively subjected to colonoscopy with an exam scheduled from 8.00 to 10.00
* Age between 18 and 75 years
* Written informed consent

Exclusion Criteria:

* Hypersensitivity and contraindications to the product under study, to the active ingredients or to any of the excipients.

Known severe renal insufficiency (Glomerular Filtration Rate (eGFR) <30 ml / min / 1.73 m2)

* Presence of known chronic inflammatory bowel disease
* Previous digestive tract surgery
* Suspected gastrointestinal perforation
* History of congestive heart failure (NYHA class III or IV)
* Severe hepatic insufficiency or impairment (in the case of Child-Pugh Class C accurate verification of the patient's condition) indicated by transaminase values greater than 3 times the maximum normal value.
* Toxic colitis or toxic megacolon
* Suspected intestinal obstruction
* Patients enrolled in colorectal cancer screening programs
* Intestinal paralysis
* Documented electrolyte disturbances (Na, Cl, K, Ca or P outside normal limits)
* Recent symptomatic acute ischemic heart disease (<6 months). Acute myocardial infarction and recent unstable angina within six months antecedents.
* Participation in a clinical trial in which an investigational drug was administered within 30 days or 5 half-lives of the study drug, whichever is longer.
* Documented state of pregnancy ascertained through positive pregnancy test

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Percentage of colonoscopies with adequate preparation | 1 day - the day of the colonoscopy
  Percentage of colonoscopies with adequate preparation (according to BBPS score ≥ 2) in each colonic segment, in patient group A vs patient group B

SECONDARY OUTCOMES:
Quantity of bubbles | 1 day - the day of the colonoscopy
  Quantity of bubbles and / or foam according to IBS, in patient group A vs patient group B
tollerability and compliance | 2 days - the day of the drug administration + the day of the colonoscopy
  Degree of acceptability, tolerability and compliance, by questionnaire, in the group of patients A vs the group of patients B

CONTACTS AND LOCATIONS:
Overall Officials: LUIGI PASQUALE, PROF, Study Chair — Societa Italiana di Endoscopia Digestiva
Locations (10):
- Italy (10):
  - Presidio Ospedaliero Sant'Ottone Frangipane, Ariano Irpino, Avellino
  - Reparto di Gastroenterologia IRRCS Saverio de Bellis, Castellana Grotte, BARI
  - SSD Endoscopia digestiva - Ospedale Manerbio, Manerbio, Brescia
  - SC Gastroenterologia Endoscopia Digestiva. Ospedale di Baggiovara, Baggiovara, Modena
  - SC Gastroenterologia ed Endoscopia Digestiva - Ospedale S. Martino, Belluno
  - Dipartimento di scienze mediche e chirurgiche, Università di Bologna - Policlinico Sant'Orsola, Bologna
  - Reparto Gastroenterologia ed Endoscopia dell'Ospedale Civile San Giovanni di Dio, Crotone
  - Servizio Centralizzato di Endoscopia Digestiva Operatoria - AOU Federico II, Napoli
  - S.S. Endoscopia Digestiva/ P.O. S. Jacopo, Pistoia
  - Chirurgia Generale AOU Policlinico Umberto I, Rome

IPD SHARING:
Plan to Share IPD: Yes
THE STUDY IS PROMOTED BY THE ITALIAN SOCIETY OF DIGESIVE ENDOSCOPY as part of research activities for the improvement of clinical practices
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: AFTER THE STUDY END NO TIME LIMIT WAS FIXED
Access Criteria: REQUEST TO THE STUDY COORDINATOR